CLINICAL TRIAL: NCT02978118
Title: Exploring Relevant Immune-based Biomarkers and Circulating Tumor Cells During Treatment With Immunotherapy in Genitourinary Malignancies
Brief Title: Exploring Relevant Immune-based Biomarkers and Circulating Tumor Cells During Treatment With Immunotherapy in Genitourinary Malignancies (CTC Immune Based Biomarkers)
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00076768
Record Dates: First submitted 2016-10-21; First posted 2016-11-30 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Renal Cell; Carcinoma, Urothelial
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Renal Cell Carcinoma: Subjects in Group A (patients with locally advanced, high grade or metastatic renal cell carcinoma starting immunotherapy) will have blood collected at baseline, at the time of a standard of care cytoreductive surgery (if applicable), 12 weeks, 24 weeks, 52 weeks and upon disease progression on treatment for analysis of peripheral blood mononuclear cells (PBMCs), circulating tumor cells (CTCs), metabolites, cytokines and angiokines. Urinary and fecal specimens will be collected at baseline, at the time of a standard of care cytoreductive surgery (if applicable), 12 weeks, 24 weeks, 52 weeks and upon disease progression. Tissue will be collected at the time of a standard of care cytoreductive surgery (if applicable).
  Interventions: Device: Immune cell and CTC detection procedures
- Group B: Urothelial Carcinoma: Subjects in Group B (patients with locally advanced, high grade or metastatic urothelial carcinoma starting immunotherapy) will have blood collected at baseline, at the time of a standard of care cytoreductive surgery (if applicable), 12 weeks, 24 weeks, 52 weeks and upon disease progression on treatment for analysis of peripheral blood mononuclear cells (PBMCs), circulating tumor cells (CTCs), metabolites, cytokines and angiokines. Urinary and fecal specimens will be collected at baseline, at the time of a standard of care cytoreductive surgery (if applicable), 12 weeks, 24 weeks, 52 weeks and upon disease progression. Tissue will be collected at the time of a standard of care cytoreductive surgery (if applicable).
  Interventions: Device: Immune cell and CTC detection procedures

INTERVENTIONS:
Device: Immune cell and CTC detection procedures — Immune cell profiling assays (in blood and archival tumor samples) and circulating tumor cell assays (in blood samples)

SUMMARY:
This pilot study purpose of this study is to describe peripheral circulating immune cell profiles at baseline and change on treatment with immune checkpoint inhibitors in renal cell carcinoma and urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Group A Renal Cell Carcinoma:

Patients will be eligible for inclusion in this study if ALL of the following criteria apply:

1. Histologically confirmed or radiological diagnosis of renal cell carcinoma. Clear cell and non-clear cell carcinoma (such as papillary, chromophobe, collecting duct, and medullary) allowed.
2. Evidence of locally advanced, high grade or metastatic disease in any site on most recent imaging scan
3. Planned initiation of treatment with any of the following:

   * Immune modulatory agent targeting any of the following: PD-1, PD-L1, CTLA-4, CD27, OX40, LAG3 or tumor infiltrating lymphocytes (TIL)
   * Immune modulatory agent consisting of any of the following: CAR-T, bispecific antibody or vaccine trial.
4. Age > 18 years.
5. Ability to understand and the willingness to sign a written informed consent document.

Group B Urothelial Carcinoma:

Patients will be eligible for inclusion in this study if ALL of the following criteria apply:

1. Histologically confirmed diagnosis of urothelial carcinoma. Non-transitional cell carcinoma (such as adenocarcinoma and squamous cell carcinoma) allowed.
2. Evidence of locally advanced, high grade or metastatic disease in any site on most recent imaging scan
3. Planned initiation of treatment with any of the following:

   * Immune modulatory agent targeting any of the following: PD-1, PD-L1, CTLA-4, CD27, OX40, LAG3 or tumor infiltrating lymphocytes (TIL)
   * Immune modulatory agent consisting of any of the following: CAR-T, bispecific antibody or vaccine trial.
4. Age > 18 years.
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. History of intercurrent or past condition that would make participation in this protocol difficult or not feasible at the discretion of the principal investigator or co-investigator(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Duke Cancer Institute Patients
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in the number of T-cells before and after treatment with immune therapies | Baseline and Disease progression (up to two years)
Change in the number of B-cells before and after treatment with immune therapies | Baseline and Disease progression (up to two years)
Change in the number of myeloid-derived suppressor cells (MDSCs) before and after treatment with immune therapies | Baseline and Disease progression (up to two years)
Change in the number of neutrophil cells before and after treatment with immune therapies | Baseline and Disease progression (up to two years)
Number of patients with detectable circulating tumor cells (CTCs) | Disease progression (up to two years)

SECONDARY OUTCOMES:
The prevalence of tumor-infiltrating lymphocytes for all subjects at baseline | Baseline
The prevalence of tumor-associated macrophages for all subjects at baseline | Baseline
The change in CTCs over time | Baseline, week 4, week 8, week 12 and progression (up to two years)
The distribution of CTCs difference scores across the ordered tumor response categories of CR, PR, SD, and PD | Disease progression (up to two years)
The change in tumor burden over time measured by RECIST | Baseline, Week 12, Progression (up to two years)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States